CLINICAL TRIAL: NCT04286932
Title: National Children's Food Consumption Survey II
Brief Title: National Children's Food Survey II
Acronym: NCFS II
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: University College Dublin (Other); Dublin Institute of Technology (Unknown)
Responsible Party: Principal Investigator, Janette Walton, Senior researcher, University College Cork
Other Study IDs: 15 F 673
Record Dates: First submitted 2017-05-15; First posted 2020-02-27 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Dietary Habits; Life Style; Body Weight
MeSH Terms: conditions — Feeding Behavior; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 5-12y

SUMMARY:
The overall objective of this project is to establish for the Republic of Ireland (ROI) a nationally representative database of food consumption in children aged 5-12 years to update 2003-04 data for this group and to complement more recent data on preschool children and adults. The survey will be comparable with existing survey data in ROI and with surveys in UK (GB & NI). The ROI database will be designed to address both nutrition and food safety issues of relevance to the development and implementation of public health policy, food safety risk assessment and to the needs of the food industry. In addition to detailed data on food consumption, data will be also be collected on body weight, lifestyle, including physical activity, determinants of food choice, urine, and composition of foods and food recipes. Food composition databases will be updated and restructured to facilitate future analyses of food ingredients, packaging materials, residues, contaminants, allergens, bioactives and microorganisms. Urine samples will be stored to facilitate future analyses nutrition and metabolic indicators, markers of food intake and for estimating exposure to food chemicals. Data will be analysed to estimate intakes of foods and nutrients and compliance with dietary recommendations, to establish the prevalence of overweight and obesity, to investigate physical activity patterns and compliance with guidelines, to identify psychological, social and attitudinal determinants of food choice and eating behaviour. Salt intake will be estimated from urine excretion. Findings will be disseminated to relevant stakeholders. The project will be carried out by a multi-disciplinary research team with strong linkages to related on-going research in food and health sciences.

ELIGIBILITY:
Inclusion Criteria:

* Attending primary school

Exclusion Criteria:

-

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Primary school children living in Ireland; 5-12y; representative of age, gender, social class, location of residence
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Food and nutrient intake of Irish children (5-12y) | Jan 2017-Dec 2019
  Participating families were asked to record detailed information on the amount and type of all foods, drinks and nutritional supplements consumed by the child over four consecutive days (including one weekend day) in a food diary. Participants were provided with digital food scales and asked to weigh as many foods as possible, including leftovers. Where foods were not weighed, researchers used age-appropriate photographic food atlases, standard portion sizes and household measures at subsequent visits to help with quantifying the amount of food consumed. Participants were encouraged to keep food packaging to provide further detail on the foods consumed. Nutrient intakes were estimated from food intakes using tables of food composition.
Anthropometry measurements of Irish children (5-12y) | Jan 2017-Dec 2019
  Physical measurements (height, weight, % body fat, and waist and hip circumference) of the children were made.
Health and Lifestyle Characteristics of Irish children (5-12y) | Jan 2017-Dec 2019
  Participants and parents/guardians completed a questionnaire on general health and lifestyle.
Food Choice Behaviour of Irish children (5-12y) | Jan 2017-Dec 2019
  Participants and parents/guardians completed questionnaires on determinants of food choice and eating behaviours for the child.
Physical Activity Measurements of Irish children (5-8y) | Jan 2017-Dec 2019
  Physical activity was estimated using the validated Child Physical Activity Questionnaire (C-PAQ) in 5-8 year olds.
Physical Activity Measurements of Irish children (9-12y) | Jan 2017-Dec 2019
  Physical activity was estimated using the the Youth Physical Activity Questionnaire (Y-PAQ) in 9-12 year olds.
Urine sample collection and analysis of Irish children (5-12y) | Jan 2017-Dec 2019
  A single first-void morning urine sample was also collected from children during the recording period to estimate sodium and potassium intake.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided